CLINICAL TRIAL: NCT06392399
Title: Cooled Radiofrequency in Comparison to Either Conventional Radiofrequency Thermocoagulation or Neurolytic Block of Ganglion Impar in the Management of Perineal Cancer Pain
Brief Title: Interventions for the Management of Perineal Cancer Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Abo eldahab Ali elden, Aya Abo Eldahab, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-2024-679
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Cancer Rectum; Cancer Vulva; Cancer Vagina
Keywords: cooled radiofrequency , conventional radiofrequency
MeSH Terms: conditions — Rectal Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional radiofrequency (Active Comparator): In this group we will use conventional radiofrequency thermocoagulation in the management of perineal cancer pain
  Interventions: Device: conventional radiofrequency
- Cooled radiofrequency (Active Comparator): In this group we will use cooled radiofrequency in the management of perineal cancer pain
  Interventions: Device: cooled radiofrequency ,
- Neurolytic block of Ganglion (Active Comparator): In this group we will use neurolysis of ganglion impar in the management of perineal cancer pain
  Interventions: Device: neurolysis of ganglion

INTERVENTIONS:
Device: cooled radiofrequency , — In Cooled RF, after placement of the introducer needle, the 18 gauge internally cooled RF electrode is used for 90 seconds at a temperature of 60°C.
  Arms: Cooled radiofrequency
Device: conventional radiofrequency — In conventional RF group lesion will be performed at 80°C for 120 seconds.
  Arms: Conventional radiofrequency
Device: neurolysis of ganglion — In neurolytic block, Once the position of the needle tip confirmed, 4 - 6 mL of 8% phenol in saline will be injected followed by 1 mL of saline to avoid the deposition of phenol within the intervertebral disc material.
  Arms: Neurolytic block of Ganglion

SUMMARY:
Pain associated with neoplasms may be of somatic, visceral, or neuropathic origin.Visceral pain or pain that is mediated by the sympathetic fibers in the perineal area associated with malignancy in the pelvis may be effectively treated with neurolysis of impar ganglion.In recent years, radiofrequency lesioning of the ganglion Impar has evolved as a novel non pharmacological technique for the management of patients suffering from intractable perineal pain.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients aged from 20-70 years old, with lower third cancer rectum, caner vulva, cancer vagina and cancer perineum.
2. The intensity of perineal pain on VAS score ≥ 5.
3. Unsatisfactory treatment with tramadol (400 mg daily) , Pregabalin (150 mg daily) or presence of side effects of tramadol as headache, dizziness, constipation, rash, sweating, dry mouth.
4. Included participants should show adequate response to diagnostic ganglion impar block , i.e. reduction of VAS pain score > 50% at least for 2 hours.

Exclusion Criteria:

1. Infection of the skin at or near site of needle puncture.
2. Coagulopathy or prolonged bleeding time.
3. Drug hypersensitivity or allergy to the studied drugs.
4. Central or peripheral neuropathy .
5. Significant organ dysfunction as respiratory , liver or renal failure.
6. Any psychiatric illness that would interfere with the perception and the assessment of pain.
7. Vertebral anomalies.

   -

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients gaining ≥ 50% reduction of their pre procedural pain at VAS Score from baseline value. | 2 hours, 24 hours,1 week, 2 weeks, 1 month, 3 months.
  Patients rate pain on a scale from 0-10, 0 being no pain and 10 being the worst pain imaginable.

SECONDARY OUTCOMES:
Total Tramadol consumption | at 2 weeks, 1 month, 2 months and 3 months' post procedural.
  we will measure consumption of tramadol either it increasing or decreasing .

OTHER OUTCOMES:
Patient's satisfaction by the Global Perceived Effect questionnaire | at baseline, 2 weeks, 1 month, 3 months.
  provides patient feedback on your empathy and relationship-building skills during consultations.

CONTACTS AND LOCATIONS:
Overall Officials: aya ali, Principal Investigator — Assiut University